CLINICAL TRIAL: NCT04096144
Title: Evaluation of Sugammadex Vs. Neostigmine in the PACU for Abdominal Surgeries
Brief Title: Comparison of Sugammadex and Neostigmine During PACU Stay
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Enrico Camporesi, Professor of Surgery, University of South Florida
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 41493
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Neuromuscular Blockade
Keywords: Post anesthesia care unit; sugammadex; neostigmine; neuromuscular reversal
MeSH Terms: interventions — Neuromuscular Blocking Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Neostigmine (Experimental): This is the standard Neuromuscular reversal drug that has been in standard care for the past thirty years. Dose: -Neostigmine: 0.03-0.07 mg/kg by intravenous route.
  Interventions: Drug: Neuromuscular Blocking Agents
- Sugammadex (Experimental): Used for Neuromuscular reversal; Sugammadex is devoid of the parasympathetic effects caused by Neostigmine.
  Dose: -Sugammadex: 2-4 mg/kg (4 mg/kg if no twitch responses after initial stimulation), intravenous route.
  Interventions: Drug: Neuromuscular Blocking Agents

INTERVENTIONS:
Drug: Neuromuscular Blocking Agents — Neuromuscular agents will be used to block muscle function for the safety and efficiency of the procedure. At the procedure's conclusion, neuromusclar agents such as Neostigmine or Sugammadex will be used to reverse the neuromuscular reversal.

SUMMARY:
Sugammadex was approved for post-operative use in the operating room (OR) and post-anesthesia recovery unit (PACU) of our quaternary facility, Tampa General Hospital. The approval came with administrative limitations: 2mg/kg dose only and for the first year its utilization was limited as replacement for up to half of Neostigmine/Glycopyrrolate use.

An MUE evaluation was completed for a retrospective chart review from March 2017 to December 2017 (10 months) to assess all cases in which patients received Sugammadex or Neostigmine. During the year of data collection, we also noted a widespread tendency to reduce the usage of narcotics.

A t-test comparison of the length of stay (LOS) in the PACU revealed a highly significant difference between the LOS in PACU for both drugs. On average, patients receiving Sugammadex were discharged from the PACU 43 minutes earlier than patients who received Neostigmine/Glycopyrrolate. The patient mix in both groups was similar, but these data were obtained retrospectively by a pharmacy chart review.

DETAILED DESCRIPTION:
Primary Objective:

* To evaluate the Length of Stay (LOS) in the PACU after a neuromuscular reversal with Sugammadex in comparison with Neostigmine/Glycopyrrolate in abdominal surgeries (hernia, gallbladder, etc.).
* Primary Endpoints: Date, Gender, Date of Procedure, Length of Procedure, Attending Anesthesiologist, Length of PACU stay (Admission and Discharge), Pain VAS score, Aldrete Score, Finger Saturation, and BP upon PACU discharge.

Study Design This is a prospective, randomized, study to evaluate the length of stay in the PACU after a neuromuscular reversal with Sugammadex in comparison with Neostigmine/Glycopyrrolate in abdominal surgeries (hernia, gallbladder surgeries, etc.) Inclusion Criteria

* 18-75 years of age
* Patients with surgeries with duration of 90-120 minutes
* ASA Patients I-III (Appendix A)
* Patients admitted to TGH for abdominal hernia repair, cholecystectomy and/or abdominal surgery as performed by Dr. Albrink
* BMI > 30 Exclusion Criteria
* <18 years of age
* ASA Patients IV and above (Appendix A)
* Patients with allergic reactions to Neostigmine+Glycopyrrolate and/or Sugammadex Patient Safety The patients enrolled in this study protocol are all in need of a general anesthetic supplemented by muscle relaxation, and able to receive rocuronium or vecuronium, the two most frequently used muscle relaxant at TGH. Both types of muscle relaxant can be reversed appropriately at the end of the surgical procedure with Bridion (sugammadex) or neostigmine in combination with Glycopyrrolate. The dose of the both reversal agents will be chosen to be equivalent for the intermediate level of neuromuscular blockade reached at the end of the surgical procedure. We have multiple year experience in using these two reversal drugs. Despite a difference in speed of onset, both drugs are commonly used in our operating room after these abdominal procedures. The reversal drugs are administered in the operating room toward the end of the procedure, when muscle paralysis of the abdominal wall is not required by the surgeon, and the anesthesiologist needs to awaken the patient and restore spontaneous ventilation. Side effects of both reversal agents might comprise especially bradycardia, usually reversed with Glyco supplementation, Other side effects and rarely allergy to the drug have been described and we are monitpring patients to maintain high safety throughout this period. The important notion is that the patient will be adequately reversed, breathing spontaneously, extubated and responding to appropriate questions before transfer to the PACU.

Methodology Consent Process All patients who are having abdominal surgeries at Tampa General Hospital (TGH) will be evaluated for study eligibility in the preoperative assessment center at TGH during their visit with the anesthesiologist. The pre-operative assessment takes place 3-7 days prior to the scheduled surgery. Patients who qualify for the study will be entered into the study during their pre-operative visit or the patient may take the consent form home to review and sign on the day of surgery. All study discussions will take place in a private exam room in the preoperative clinic. All subjects will be given the opportunity to ask questions. If the investigator feels that the subject understands the research parameters and the subject is willing to sign the consent form, the patient will be enrolled in the study. On the day of the surgical procedure, the study subject will present to the surgical prep unit. It is here that the subject will be re-evaluated for willingness to participate. Any additional questions will be answered prior to surgery.

Patients will be sedated with propofol and will be maintained with Sevoflourane. Rocuronium will be used to relax the muscles. Reversal will be administered with two or more twitches, according to the TOF monitor.

Screening & Baseline Visit After the patient signs the consent form, patient demographics and medical history will be collected from the medical record. A clinical examination, including vital signs (blood pressure, heart rate, and respiratory rate); physical measurements (body weight and body height) and physical examination will be completed.

Surgery Fifty subjects will be enrolled in the study. Fifty randomized envelopes will be used to make the selection of the drug on the day of surgery. If the surgery is the first case of the day, the selection will be made the afternoon prior to the day of surgery. The drugs will be stored and utilized in the OR as part of standard practice. If the dose for reversal is administered more than once, the patient will be immediately withdrawn from the study.

Monitoring in the PACU After the patient has completed the surgery, he/she will be extubated and transferred to the PACU where vital signs are monitored every 3-5 minutes. Patients will be discharged from the PACU by a PACU nurse under the guidance of the providing anesthesiologist.

Statistical Analysis Sample Size: Sixty subjects will be enrolled in the study, to account for patient dropout. Sample size selection is based on referral from the Co-Investigator, Dr. Michael Albrink. We hope to use data from this study to develop a larger study including sample size determination with power analysis using our findings from this study.

Data Analysis: The length of stay (LOS), Aldrete scores, as well as Pain VAS scores will be compared for each respective drug. Univariate analyses will be used for distribution (ranges of values, frequency distribution), central tendency (mean, median, mode), and dispersion (range, standard deviation).

Data Safety Monitoring:

Enrico M. Camporesi, M.D. and Maha Balouch, B.A. will ensure the integrity of the data collected by verifying the accuracy of the data recorded against the medical records. Monitoring will occur on a weekly basis. Any action resulting in a temporary or permanent suspension of the study will be reported to the IRB. The collection of personal patient information will be limited to the amount necessary to achieve the aims of the research, so that no unneeded sensitive information is being collected. Only study personnel will collect data. Hard copy documents will be retained for the duration of the study until data entry. All hard copy documents will be kept in a locked cabinet in the research coordinator's office. All electronic data will be recorded in a password protected Excel spreadsheet and data analysis will be conducted using de-identified data in SPSS statistical software. All hard copy documents will be shredded within five years after completion of the study.

Risks Both of these drugs may cause post-operative nausea and vomiting (PONV). Benefits Although the patient may not receive any benefit from participating in this study, medical science and future patients may benefit from his/her participation.

Study Plan The study will be conducted over 6-8 months. Patients will only be involved in the study while they are in the Post-Anesthesia Care Unit.

Timeline:

* 4-5 months: consenting and enrolling patients; data collection
* 2-3 months: data analysis and writing of abstracts/paper Publication Plan We plan on submitting abstracts to the American Society of Anesthesiologists (ASA) Meeting and the Society of Anesthesia and Sleep Medicine (SASM) Meeting. Eventually, we would like to publish our work in a peer-reviewed journal.

A description of this clinical trial will be available on www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Patients with surgeries with duration of 90-120 minutes
* ASA Patients I-III (Appendix A)
* Patients admitted to TGH for abdominal hernia repair, cholecystectomy and/or abdominal surgery as performed by Dr. Albrink
* BMI > 30

Exclusion Criteria:

* <18 years of age
* ASA Patients IV and above (Appendix A)
* Patients with allergic reactions to Neostigmine+Glycopyrrolate and/or Sugammadex

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Length of Post Anesthesia Care Unit (PACU) stay | 6 months
  Time spent in the recovery room (PACU).
Pain (Visual Analog Scale) VAS scores | 6 months
  Evaluation of the level of pain
Aldrete Score | 6 months
  Evaluation of level of alertness of the patient at the conclusion of PACU stay for discharge.
Pulse Oximetry | 6 months
  Finger Saturation
Blood Pressure upon PACU discharge | 6 months
  Evaluation of Blood Pressure at the conclusion of PACU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Camporesi, MD, Principal Investigator — TEAMHealth Anesthesia/Tampa General Hospital; Maha Balouch, MA, Study Chair — TEAMHealth Anesthesia/Tampa General Hospital; Michael Albrink, MD, Principal Investigator — Tampa General Hospital
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Enten G, Albrink M, Deng J, Melloni G, Camporesi EM, & Mangar D. Sugammadex Administration Shortens Reversal Times but not OR Turnover Times. Case Studies in Surgery. 2019 Jul;5(1): 27.
- [Background] Presented at 2019 American Society of Anesthesiologists meeting: Mangar D, Pease S, Guzman S, Abowali H, Balouch M, & Camporesi EM. PACU Length of Stay after Neuromuscular Blocker Reversal with Sugammadex. Orlando, FL.